CLINICAL TRIAL: NCT03001089
Title: Impact of the Administration of Fludrocortisone on Fluid and Electrolyte Balance in Very Premature Infants: Pilot Study
Brief Title: Impact of the Administration of Fludrocortisone in Very Premature Infants
Acronym: MINIPREM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P150905
Record Dates: First submitted 2016-12-12; First posted 2016-12-22 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Partial Mineralocorticoid Deficiency
Keywords: Neonatology; Endocrinology
MeSH Terms: interventions — Fludrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fludrocortisone 10 µg tablets (Active Comparator): Oral Fludrocortisone (enteral) at a dose of 10 mcg 2 times daily (every 12 hours) for 8 days from day 1 (first administration between H24 and H30, and then every 12 hours) until day 8.
  Interventions: Drug: Oral Fludrocortisone (enteral)
- placebo oral tablet (Placebo Comparator): Oral placebo (enteral) at a dose of 10 mcg 2 times daily (every 12 hours) for 8 days from day 1 (first administration between H24 and H30, and then every 12 hours) until day 8.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Oral Fludrocortisone (enteral) — Oral Fludrocortisone (enteral) at a dose of 10 mcg 2 times daily (every 12 hours) for 8 days from day 1 (first administration between H24 and H30, and then every 12 hours) until day 8.
  Arms: Fludrocortisone 10 µg tablets
Drug: Placebo Oral Tablet — oral placebo (enteral) at a dose of 10 mcg 2 times daily (every 12 hours) for 8 days from day 1 (first administration between H24 and H30, and then every 12 hours) until day 8.
  Arms: placebo oral tablet

SUMMARY:
Water and electrolytic homeostasis is remarkably controlled by the mineralocorticoid pathway (renin-angiotensin-aldosterone system acting on the renal tubule). However, the neonatal period in humans is characterized by a reduced ability of the kidney to ensure normal functions of urine concentration and maintenance of sodium and water balance. This renal functional immaturity, is associated in the very premature infants (VPT) (born <32 weeks of amenorrhea (SA)) to an immaturity of the adrenal responsible for a default of aldosterone biosynthesis . This relative aldosterone deficiency induces difficulties for VPT to adapt to extra-uterine life when maintaining a positive sodium balance is essential for postnatal growth. The improvement of perinatal care (antenatal corticosteroids maturation, ventilation techniques and use of surfactant) have increased the survival of these children . Nevertheless, extreme prematurity (less than 32 weeks), which concerns nearly 2% of live births in France, remains associated with neurodevelopmental sequelae in nearly 40% of children at 5 years .

Secondary hydroelectrolytic disorders with transient mineralocorticoid adrenal insufficiency is probably one of the factors responsible of these neurological deleterious outcomes as well as the occurrence of other complications (bronchopulmonary dysplasia, enterocolitis necrotizing) of extreme prematurity. Indeed, aside from the administration of antenatal steroids to induce maturation, the prevention of postnatal dehydration reduces the risk of intracranial hemorrhage in that population. However, high fluid intake are associated with an increased incidence of patent ductus arteriosus, of bronchopulmonary dysplasia and necrotizing enterocolitis. This necessitates the evaluation of preventive measures to avoid such fluid and electrolyte imbalances by a pharmacological approach based on mineralocorticoid administration in very premature infants, due to the relative aldosterone deficiency identified in this population.

DETAILED DESCRIPTION:
Extreme prematurity affects about 2% of births per year in France and is subject to a significant morbidity and mortality. It is likely that the fluid and electrolyte imbalances associated with mineralocorticoid adrenal insufficiency transient observed in this population of vulnerable newborns contribute to the occurrence of complications that will influence the prognosis medium and long term these children. The expected impact of our pilot study is a direct benefit to the patient, with reduced kidney soda losses from the 3rd day of life and throughout the first week of life (assessed by a non-invasive method: urine collection to compress and measurement of urinary Na / creatinine). This physiological approach (substitution of the deficient hormone) allow better control of sodium and water balance. This could limit a number of common complications of extreme prematurity, occurring in the first weeks of life, such as patent ductus arteriosus, intra-ventricular hemorrhage and bronchopulmonary dysplasia.

The administration of glucocorticoids during the postnatal period (with action both glucocorticoid and mineralocorticoid) enables a reduction in the incidence of bronchopulmonary dysplasia severe. However, such treatment is associated with an increased incidence of neurodevelopmental effects related to activation of the glucocorticoid pathway. Using a specific mineralocorticoid agonist should preserve the beneficial effects without the adverse effects observed. The results of this pilot study will in a second time to consider a clinical trial Phase III national or international evaluating the significant reduction of these complications after substitution by Fludrocortisone the first week of life in the great premature. These results should have a major medical and economic impact. Indeed, neonatal morbidity indicators (intraventricular hemorrhage, patent ductus arteriosus, bronchopulmonary dysplasia and enterocolitis necrotizing) are associated with the subsequent development of neurodevelopmental sequelae (cerebral palsy and / or cognitive impairment) at the age of two and five years.

ELIGIBILITY:
Inclusion Criteria:

* Very premature newborns defined by a gestational age <32 and ≥ 26 gestational weeks
* Eutrophic: birth weight between the 10th and 90th percentile of the French reference curves
* Absence of malformations or chromosomal abnormality identified
* Lack of adrenal, pituitary or gonadal diseases diagnosed prior birth
* Lack of participation in another research protocol
* "Inborn": born and hospitalized in the four neonatology departments participating in the study
* Informed consent of the holders of parental authority

Exclusion criteria:

* Maternal treatment prior to pregnancy: systemic or inhaled corticosteroids, hormone therapy for adrenal or pituitary insufficiency, antihypertensive treatment (calcium channel blockers, beta blockers, angiotensin)
* Lack or incomplete treatment of antenatal glucocorticoids (betamethasone)

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Urinary sodium loss evaluated by the urinary ratio Na / creatinine | day 3 (when urinary sodium losses are at their highest in very premature infants)
  Measurement of Na / urinary creatinine ratio at day 3 (evaluating the efficacity of Fludrocortisone action on the kidney by lowering sodium losses, that are very high in very premature infants) by collection of a urinary spot collected on a gauze compress, placed in the diaper of the newborn.

SECONDARY OUTCOMES:
Urinary sodium loss evaluated by the urinary ratio Na / creatinine | day1, day5, day8, day10 and day15
  Measurement of Na / urinary creatinine ratio at day 1, 5, 8, 10 and 15 (evaluating the efficacity of Fludrocortisone action on the kidney by lowering sodium losses, that are very high in very premature infants) by collection of a urinary spot collected on a gauze compress, placed in the diaper of the newborn.
urinary sodium and potassium concentrations | day1,day3, day5, day8, day10 and day15
plasma sodium and potassium concentrations | day1, day3, day8 et day15
plasma renin concentrations | day1, day3, day8 et day15
Number of blood tests | day1,day3, day5, day8, day10 and day15
Neonatal complications | up to 36 post-conceptional weeks (PCW)
Patent ductus arteriosus (diagnosed by ultrasound) | Between day2 and day5 and between day7 and day15
Presence of intraventricular hemorrhage (diagnosed by ultrasound) | between day2 and day5, and between day7 and day15, and at the age of 36 PCW
Oxygen inspired fraction (FiO2) | At Day 28 and 36 PCW
Blood pressure | From day1 to day8, at day10, at day15, at one month, three month, six month, twelve month and at 36 PCW
urinary dosage of aldosterone and cortisol | At one month, three month, six month and twelve month.
urinary index (Aldosterone/Nau) | day3, day8 and day15
number of days of invasive and non invasive ventilation | At Day 28 and 36 PCW
weight newborns | from day1 to day 8, at day 10 and day 15and at 36 PCW

CONTACTS AND LOCATIONS:
Overall Officials: Martinerie Laetitia, PHD, Principal Investigator — APHP
Locations (1):
- Hôpital Robert Debré, Paris, France

IPD SHARING:
Plan to Share IPD: No